CLINICAL TRIAL: NCT06513260
Title: Evaluation of the Effect of Virtual Reality Distraction on Controlling Dental Anxiety During the Surgical Extraction of Impacted Lower Third Molar Teeth
Brief Title: Effect of Virtual Reality Distraction on Anxiety Control During Impacted Molar Tooth Surgery
Status: Completed | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, EDA İZGİ, Assistant Professor Doctor, Kutahya Health Sciences University
Other Study IDs: KutahyaHSU/Edaİzgi/001
Record Dates: First submitted 2024-07-10; First posted 2024-07-22 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Dental Anxiety; Impact Molar; Virtual Reality
Keywords: Dental Anxiety; Impact Molar; Virtual Reality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Virtual reality application: Application of virtual reality glasses during surgical extraction of impacted lower third molars.
  Interventions: Procedure: Surgical extraction of impacted lower third molars.
- No application: No application of virtual reality glasses during surgical extraction of impacted lower third molars.
  Interventions: Procedure: Surgical extraction of impacted lower third molars.

INTERVENTIONS:
Procedure: Surgical extraction of impacted lower third molars. — Surgical extraction of impacted mandibular third molars in the mesioangular position, according to the Tetsch and Wagner classification

SUMMARY:
The goal of this clinical trial is to investigate the effectiveness of virtual reality distraction therapy using virtual reality glasses in reducing dental anxiety during the surgical extraction of impacted lower third molar teeth.The main questions it aims to answer are:

* Is the use of the virtual reality distraction during the procedure effective on perceived pain and anxiety?
* Evaluation of the effectiveness of the virtual reality distraction based on initial anxiety test scores.
* Does the use of the virtual reality headset cause difficulties for the clinician in performing the procedure?

Patients will undergo anxiety tests before surgery.

Pre-operative vital signs will be recorded.

The procedure will be performed either with or without virtual reality glasses, according to the randomly assigned groups.

Post-operative vital signs will be recorded.

At the end of the procedure, all patients will undergo anxiety tests and verbal rating scales.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* Being systemically healthy
* Needing surgical extraction treatment of impacted lower third molar (in mesioangular position according to Tetsch and Wagner Classification)
* Having a score of 11 or higher on the dental anxiety scale

Exclusion Criteria:

* History of seizures or convulsive disorders
* Balance disorders such as nystagmus or vertigo
* Use of psychotropic medications
* Undergoing treatment for anxiety
* Patients with psychiatric disorders
* Presence of dermatological lesions, especially around the face and eyes
* Presence of any lesion in the eye that would prevent the use of virtual reality
* Presence of systemic diseases and medication use contraindicating surgical extraction of impacted teeth

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: - Healthy volunteers
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Modified Dental Anxiety Scale Scores | Baseline
  In patients with and without the use of virtual reality glasses, the dental anxiety scale and verbal rating scales evaluating their experience during the treatment will be applied.
Heart rate measurements | During the operation
  In patients with and without the use of virtual reality glasses, heart rate will be monitored before, during, and after the treatment.
Blood pressure measurements | During the operation
  In patients with and without the use of virtual reality glasses, blood pressure will be monitored before, during, and after the treatment.
Oxygen saturation measurements | During the operation
  In patients with and without the use of virtual reality glasses, saturation will be monitored before, during, and after the treatment.

SECONDARY OUTCOMES:
Dentist feedback | Baseline
  Verbal rating scales will be applied to the dentist to evaluate the potential difficulties associated with the use of virtual reality distraction.

CONTACTS AND LOCATIONS:
Overall Officials: Eda İzgi, Principal Investigator — Kutahya University of Health Sciences
Locations (1):
- Kütahya Health Science University, Kütahya, Turkey (Türkiye)